CLINICAL TRIAL: NCT02561949
Title: Adapting Mental Health Interventions for War-Affected Youth Through Employment Programs in Sierra Leone
Brief Title: Adapting Mental Health Interventions for War-Affected Youth Through Employment Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: Caritas Freetown (Other); World Bank (Other); The City College of New York (Other)
Responsible Party: Principal Investigator, Theresa Betancourt, Salem Professor in Global Practice, Boston College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0603-04
Record Dates: First submitted 2015-09-25; First posted 2015-09-28 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Anxiety Disorder/Anxiety State; Depressive Disorder/Psychology; Social Problems/Psychology; Violence, Non-accidental
Keywords: Depression/therapy; Developing Countries; Interpersonal Relations; Life Change Events; Psychotherapy, group; Resilience, Psychological; Sierra Leone; Survivors/psychology; Social Adjustment; Social Behavior; War
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Depression; Social Adjustment; Social Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- YRI + Employment Program (Experimental): Immediately following enrollment participants will complete the YRI intervention, followed by an income generating activity program.
  Interventions: Behavioral: YRI; Other: Income generating activity program
- Employment Program (Experimental): Immediately following enrollment participants will complete an income generating activity program.
  Interventions: Other: Income generating activity program

INTERVENTIONS:
Behavioral: YRI — Youth Readiness Intervention (YRI) is an innovative, evidence-based mental health intervention to address co-morbid difficulties with externalizing problems (anger/emotion dysregulation) and internalizing problems (hopelessness/anxiety) among violence-affected youth. YRI methodology draws on evidence-based treatment elements commonly used in both cognitive-behavioral intervention and group interpersonal therapy. YRI has cross-cutting efficacy across a range of mental health conditions common in violence-affected youth. YRI will be delivered in 12 sessions over the course of 3 months.
  Other Names: Youth Readiness Intervention
  Arms: YRI + Employment Program
Other: Income generating activity program — Income generating activity programming will be carried out by GOAL in partnership with St. George's foundation through use of their current funding. GOAL focuses on supporting people in need by providing healthcare resources, advocating and advancing child protection practices and policies, and administering livelihood programs to empower them improve their lives in a sustainable manner. The St. George's Foundation's addresses child welfare concerns by actively reaching out to homeless and orphaned children. The program is 4 months in length and consists of skills training, soft skills development (primarily in numeracy and literacy), and a cash transfer of $200.

SUMMARY:
The research will first examine data obtained from YRI participants to investigate effects of the group sessions on psychosocial functioning outcomes in youth aged 15 - 24. The research also intends to examine whether youth participating in YRI and complementary income generating activities will fare better than an employment only control group. Finally, the research intends to examine whether utilizing lay health workers are a is cost-effective and scalable method for addressing mental health concerns.

The research will investigate the following hypotheses:

1. Participants who are exposed to YRI will demonstrate greater reduction in mental health and behavioral problems than participants who are waitlisted for YRI over the same period; emotion regulation will operate as a major mechanism of YRI improvements; high comorbidity will be a treatment modifier;
2. Improvements in mental health and functioning due to YRI will lead to (mediate) greater employment outcomes and superior economic self-sufficiency over time; and
3. Homelessness, orphanhood, young parenthood, and high problems in emotion regulation co-morbid with other mental health conditions will be major moderators lessening the effectiveness of YRI.
4. Lay and trained practitioners at agencies participating in the combined mental health-employment program will demonstrate high fidelity to evidence-based treatment components and that good satisfaction, social support, and professional exchange of evidence-based practices will emerge.

DETAILED DESCRIPTION:
In Sierra Leone, a dangerous gap remains between long-term psychosocial needs and adequate services. As youth affected by the war begin to enter adulthood, they face new challenges including unemployment, interrupted education, the need to support families, marginalization and stigma, as well as the remaining psychological effects of exposure to war. Healthy social integration is critical to the long-term wellbeing of this generation, but the evidence base on effective interventions to improve skills and self-efficacy is severely limited. Despite the high burden of mental health problems among war-affected youth in Sub-Saharan Africa, few empirically-supported behavioral treatments (ESBTs) or evidence-based interventions have been implemented in this region. This study stands to make an important contribution to knowledge on effective and culturally-sensitive mental health services that can be implemented in settings fraught by multiple hardships, including war, poverty, low educational attainment, and other hardships.

This exploratory randomized control study of youth aged 15-24 comparing outcomes among youth participating in YRI proceeding enrollment in an income generating activity program (YRI + EP) to a control group that participates only in income generating activity programs (EP). This study is not fully powered to detect differences between groups and is instead a test of the intervention feasibility and acceptability, with quantitative participant assessments occurring at baseline, 3-months, 6-months, and 12-months with respect to employment related measures, and participant and interventionists interviews to elucidate mechanisms by which the intervention was more or less successful.

The YRI is an evidence-based group intervention developed in 2010 to address key emotional, behavioral, and functioning difficulties identified by the PI's prior longitudinal study of war-affected youth. The YRI has three overarching goals: (1) To improve interpersonal and community relationships through work with youth and community members; (2) To help vulnerable youth develop skills in emotional regulation, problem-solving, and interpersonal interactions necessary to be successful members of their communities; (3) To promote the healthy integration of difficult memories for youth who experience difficulties due to traumatic exposure. Primary mental health outcomes include decreased anxiety, hostility, and depression, and increased pro-social attitudes, as measured by the Oxford Refugee Studies Psychosocial Adjustment Scale and the African Youth Psychosocial Assessment. During this study YRI will be delivered by trained counselors,

Income generating activity programming will be carried out by GOAL and their partner St. George's Foundation through use of their current grant funding. GOAL focuses on supporting people in need by providing healthcare resources, advocating and advancing child protection practices and policies, and administering livelihood programs to empower them improve their lives in a sustainable manner. The St. George's Foundation's addresses child welfare concerns by actively reaching out to homeless and orphaned children. Their already existing employment program is 4 months in length and consists of skills training, soft skills development (primarily in numeracy and literacy), and a cash transfer of $200. The employment intervention is carried out by social workers and counselors, who have been trained to support delivery of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be between the ages 15-24 (UN definition of youth);
2. Participants must have an elevated score on internalizing (depression/anxiety) or externalizing (aggression/ hostility) on a measure validated for use in Sierra Leone;
3. Participants must report some impairment in daily functioning as a result of emotional or behavior problems based on a series of questions adapted from the WHODAS; and
4. Participants must neither be enrolled in school nor have gainful employment of 20 or more hours of work per week over the past four weeks.

Exclusion Criteria:

1. Participant fails to meet the age requirements;
2. Participant is either currently enrolled in school or has gainful employment of 20 hours or more of work per week over the past four weeks;
3. Participant is not in favor of joining an employment program;
4. Participants does not have an elevated score on internalizing (depression/anxiety) or externalizing (aggression/ hostility) on a measure validated for use in Sierra Leone;
5. Participant does not report some impairment in daily functioning as a result of emotional or behavior problems based on a series of questions adapted from the WHODAS;
6. Participant identified by clinical staff as: (a) experiencing suicidality, or (b) psychosis.

Participants at risk of harm to themselves or others, as well as those requiring treatment beyond the scope of YRI will be referred to local mental health or social work treatment facilitates as appropriate.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in % of youth with improved health outcomes | Baseline, 3 months, 6 months, and 12 months
  The percent of youth with improved mental health and daily functioning will be measured through a quantitative assessment battery including measurements from the Hopkins Symptoms Checklist, Oxford Measure of Psychosocial Adjustment, Ways of Coping Questionnaire, UCLA Traumatic Stress Disorder Reaction Index, World Health Organization Disability Adjustment Scale, Difficulties in Emotion Regulation Scale.

SECONDARY OUTCOMES:
YRI Fidelity Protocol | 3 months
  Feedback will be gained on the more or less successful programmatic mechanisms and the intervention quality and sustainability through semi-structured qualitative exit interviews with interventionists and youth.
Change in knowledge, attitudes, and behaviors of youth around employment and access to employment services. | 6 months
  Supervisors will assess youth on attendance, workplace performance, economic self-sufficiency, financial consumption/expenditures, savings and employment-related behaviors (supervisors will be interviewed about each young person blind to their group assignment).

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Betancourt, ScD, MA, Principal Investigator — Harvard University T.H. Chan School of Public Health
Locations (1):
- CARITAS, Freetown, Sierra Leone